CLINICAL TRIAL: NCT06701630
Title: Functional and Behavioural Scales Validation in Italian.
Brief Title: Italian Adaptation and Validation of Functional and Behavioural Scales for Subjective Cognitive Decline, Mild Cognitive Impairment and Mild Dementia.
Acronym: ITA-VALI-DEM
Status: Recruiting | Type: Observational
Sponsor: Casa di Cura IGEA (Other)
Responsible Party: Principal Investigator, Sabrina Guzzetti, Psychologist, principal investigator, Casa di Cura IGEA
Other Study IDs: 4920_11.09.2024_P_bis
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Neurologically Unimpaired Elderly Participants; Subjective Cognitive Decline (SCD); Mild Cognitive Impairment (MCI); Major Neurocognitive Disorder
Keywords: BADL and IADL; FAQ scale; ECog; NPI-Q; Italian adaptation; Validation; Functional and behavioral scales
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Neurologically unimpaired participants: i) Age ≥ 60 years; ii) Availability of an informant/caregiver, able to judge their functional abilities; iii) Normal performance on the Mini Mental State Examination (Folstein et al. 1975; Foderaro et al., 2022).
- Subjective Cognitive Decline (SCD): i) Age ≥ 60 years; ii) Availability of an informant/caregiver, able to judge their functional abilities.
  iii) Conditions consistent with Subjective Cognitive Decline according to Jessen et al. (2014)
- Mild Cognitive Impairment (MCI): i) Age ≥ 60 years; ii) Availability of an informant/caregiver, able to judge their functional abilities.
  iii) Conditions consistent with Mild Cognitive Impairment according to Winblad et al. (2004)
- Major Neurocognitive Disorder: i) Age ≥ 60 years; ii) Availability of an informant/caregiver, able to judge their functional abilities iii) Conditions consistent with a Mild Major Neurocognitive Disorder according to DSM-5-TR (APA, 2022).

SUMMARY:
The first aim of the observational study is the translation, cross-cultural adaptation and validation of functional and behavioral scales used in the diagnosis of neurodegenerative diseases, for which a formal version in Italian is not available at present. In particular, the study includes the following functional and behavioral scales: the Katz's index (Basic Activities of Daily Living, BADL), the Lawton and Brody's scale (Instrumental Activities of Daily Living, IADL), the Everyday Cognition questionnaire (E-Cog), the Neuropsychiatric Inventory Questionnaire (NPI-Q) for assessing the Behavioral and Psychological Symptoms of Dementia. Furthermore, a modified Italian version of the Functional Activities Questionnaire (FAQ), which integrates and updates the content of the original items (e.g., addressing the use of technologies, M-FAQ) will be used in the validation study.

The second aim is to evaluate the psychometric properties of the M-FAQ, the ECog, and the NPI-Q in terms of reliability and validity.

The third aim is to apply a Receiver Operating Characteristic (ROC) curve analysis to identify cut-offs of IADL, M-FAQ and ECOG to discriminate between different clinical groups (i.e., neurologically unimpaired elderly; Subjective Cognitive Decline, SCD; Mild Cognitive Impairment, MCI; mild Alzheimer's Disease, AD).

Neurologically unimpaired elderly participants (over 60 years old) and participants with SCD, MCI, mild AD, and their caregivers/informants will undergo: i) administration of the translated versions of the scales; ii) administration of a Cognitive Reserve questionnaire. For SCD, MCI and AD participants, data from the clinical neuropsychological evaluation will also be collected, while paper-and-pencil psychometric tests to assess global cognitive functioning (Mini Mental State Examination) and logical-abstract reasoning (Raven's Colored Matrices) will be administered to the neurologically unimpaired participants.

DETAILED DESCRIPTION:
Background Increasing aging in high-income countries, linked to increased life expectancy and declining birth rates, is accompanied by an exponential increase of dementia.

While the use of psychometric cognitive tests validated in different clinical populations is commonly used in clinical practice, there is a relative lack of validated Italian-language tools to assess functional autonomy abilities and detect the presence of neuropsychiatric symptoms, even though these are essential aspects for diagnostic, prognostic, and preventive purposes.

The assessment of functional indepedence is particularly important in the diagnosis of Mild Cognitive Impairment (MCI), where the presence of substantially intact or minimally impaired functional abilities is not easy to operationalize and measure, although it has significant relevance especially in the differential diagnosis with overt mild dementia. Currently, the functional scales most used in clinical settings are the Basic Activities of Daily Living scale (BADL), the Instrumental Activities of Daily Living scale (IADL) and the Functional Activities Questionnaire (FAQ). However, the Italian versions of these tools are informal. The group of Farias and colleagues (2008) has more recently developed a new assessment tool, the Everyday Cognition questionnaire (ECog), with a focus on functional changes in specific cognitive domains (memory, language, visuospatial skills, and executive functions).

The Neuropsychiatric Inventory (NPI) is one of the most widely used tools for assessing the Behavioral and Psychological Symptoms of Dementia (BPSD) in research, covering a wide range of neuropsychiatric symptoms. In 2000, a questionnaire form was published, the Neuropsychiatric Inventory Questionnaire (NPI-Q), which is more suitable for use in routine clinical practice and has been validated in several countries, but not in Italian.

Study design According to a power analysis, 300 neurologically unimpaired elderly participants and 90 participants, divided into Subjective Cognitive Decline (SCD), Mild Cognitive Impairment (MCI) and mild Alzheimer's Disease (AD), will participate in the study.

Inclusion criteria:

For all groups: i) Age ≥ 60 years; ii) Availability of an informant/caregiver, able to judge their functional abilities.

For neurologically unimpaired elderly: i) Normal performance on the Mini Mental State Examination.

For clinical groups: conditions consistent with:

* Subjective Cognitive Decline;
* Mild Cognitive Impairment;
* Mild Major Neurocognitive Disorder. Exclusion criteria
* Other neurological or psychiatric conditions that may explain the presence of cognitive difficulties and refusal or inability to sign informed consent.

Methods Participants and their caregivers/informants will undergo: i) Detailed information of the purpose and modalities of the study, verification of eligibility criteria, signing of informed consent; ii) Collection of demographic and anamnestic data; iii) Administration of the translated versions of the functional rating scales and NPI-q; iiii) Administration of a Cognitive Reserve questionnaire (e.g., Cognitive Reserve Index questionnaire).

For SCD, MCI and AD participants, data from the neuropsychological evaluation clinically performed will also be collected.

Two paper-and-pencil psychometric tests will be administered to neurologically unimpaired participants, to assess global cognitive functioning (Mini Mental State Examination) and logical-abstract reasoning (Raven's Colored Matrices).

Each functional scale will be administered both in the self-report version, in which the participant will provide responses relative to his or her own functioning, and in the informant version, in which the informant or caregiver will be asked to give a rating to his or her relative or friend's functioning in daily activities. The NPI-Q will be administered only to the informant.

Socio-demographic information (age, gender, manual laterality, education, and cognitive reserve assessed through specific questionnaires, e.g., CRI-Q) will be collected from all participants.

A pilot version of each translated scale will be administered, as a semi-structured interview, to about 20 participants and their informants, in order to obtain a final version for each tool to be used in the validation study.

Statistical analysis The distribution of the responses provided by the four clinical groups to the different items of the functional scales (ADL, IADL, M-FAQ and ECog) and the NPI-Q questionnaire will be analyzed to detect the presence of any ceiling and floor effects. The degree of agreement between the self-administered version and the informant version in each tool will be assessed. Cronbach's Alpha coefficient will be employed to analyze the internal consistency of ECOG, M-FAQ and NPI-Q. Convergent validity between functional scales will be calculated.

A confirmatory factor analysis will be employed to examine the factorial structure of the ECog compared to the original version.

Discriminant validity will be assessed by comparing M-FAQ and ECOG by the four scores in different clinical groups through logistic regression models.

Finally, a Receiver Operating Characteristic (ROC) curve analysis will finally be applied to identify cut-offs of IADL, M-FAQ, and ECOG to discriminate among the different clinical groups.

Expected results Italian versions of functional and behavioral scales will be obtained, according to a rigorous cross-cultural adaptation procedure, and overcoming divergences between the available Italian informal versions.

The study will also make available a modified version of the Functional Activities Questionnaire (M-FAQ) that integrates and updates the original items.

Pre-clinical and clinical validation of the tools included in the study will improve early diagnosis and longitudinal monitoring overtime.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Availability of an informant/caregiver, able to judge their functional abilities.

For neurologically unimpaired elderly:

- Normal performance on the Mini Mental State Examination (Folstein et al. 1975; Foderaro et al., 2022).

For clinical groups: Conditions consistent with:

* Subjective Cognitive Decline (Jessen et al., 2014)
* Mild Cognitive Impairment (Winblad et al., 2004)
* Mild Major Neurocognitive Disorder according (DSM-5-TR, APA, 2022).

Exclusion Criteria:

* Refusal or inability to sign informed consent;
* For the clinical groups: other neurological or psychiatric conditions that may explain the presence of cognitive difficulties.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll neurologically unimpaired participants and participants with SCD, MCI, and mild dementia referred to the Center for Cognitive Disorders and Dementia.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Everyday Cognition questionnaire score | From enrollment to the end of the assessment (1 day)
  The tool assesses functional changes in specific cognitive domains (memory, language, visuospatial skills, and executive functions).

SECONDARY OUTCOMES:
Basic Activities of Daily Living (BADL) score | From enrollment to the end of the assessment (1 day)
  The tool assesses functional autonomy in simple everyday activities.
Instrumental Activities of Daily Living (IADL) score | From enrollment to the end of the assessment (1 day)
  The tool assesses functional autonomy in instrumental everyday activities.
Functional Activities Questionnaire (FAQ) score | From enrollment to the end of the assessment (1 day)
  The tool assesses functional autonomy in complex everyday activities
Neuropsychiatric Inventory Questionnaire (NPI-Q) score | From enrollment to the end of the assessment (1 day)
  The tool assesses Behavioral and Psychological Symptoms of Dementia (BPSD) , covering a wide range of neuropsychiatric symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Guzzetti, Principal Investigator — Casa di Cura IGEA, Milan, Italy
Locations (1):
- Casa di Cura Igea, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foderaro G, Isella V, Mazzone A, Biglia E, Di Gangi M, Pasotti F, Sansotera F, Grobberio M, Raimondi V, Mapelli C, Ferri F, Impagnatiello V, Ferrarese C, Appollonio IM. Brand new norms for a good old test: Northern Italy normative study of MiniMental State Examination. Neurol Sci. 2022 May;43(5):3053-3063. doi: 10.1007/s10072-021-05845-4. Epub 2022 Jan 6. PMID 34989910
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] American Psychiatric Association. (2022). Diagnostic and statistical manual of mental disorders (5th ed., text rev.). https://doi.org/10.1176/appi.books.9780890425787
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Jessen F, Amariglio RE, van Boxtel M, Breteler M, Ceccaldi M, Chetelat G, Dubois B, Dufouil C, Ellis KA, van der Flier WM, Glodzik L, van Harten AC, de Leon MJ, McHugh P, Mielke MM, Molinuevo JL, Mosconi L, Osorio RS, Perrotin A, Petersen RC, Rabin LA, Rami L, Reisberg B, Rentz DM, Sachdev PS, de la Sayette V, Saykin AJ, Scheltens P, Shulman MB, Slavin MJ, Sperling RA, Stewart R, Uspenskaya O, Vellas B, Visser PJ, Wagner M; Subjective Cognitive Decline Initiative (SCD-I) Working Group. A conceptual framework for research on subjective cognitive decline in preclinical Alzheimer's disease. Alzheimers Dement. 2014 Nov;10(6):844-52. doi: 10.1016/j.jalz.2014.01.001. Epub 2014 May 3. PMID 24798886
- [Background] Nucci M, Mapelli D, Mondini S. Cognitive Reserve Index questionnaire (CRIq): a new instrument for measuring cognitive reserve. Aging Clin Exp Res. 2012 Jun;24(3):218-26. doi: 10.3275/7800. Epub 2011 Jun 20. PMID 21691143
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Farias ST, Mungas D, Reed BR, Cahn-Weiner D, Jagust W, Baynes K, Decarli C. The measurement of everyday cognition (ECog): scale development and psychometric properties. Neuropsychology. 2008 Jul;22(4):531-44. doi: 10.1037/0894-4105.22.4.531. PMID 18590364
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249